CLINICAL TRIAL: NCT00119509
Title: HPV DNA Testing Versus Conventional Management for Women With Minor Atypia on Pap Smear: Psychosocial and Quality of Life Outcomes and Development of a Decision Analytic Model
Brief Title: The IMAP Study Improving Management of Mildly Abnormal Pap Smears
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Family Planning Association New South Wales (Other Government)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 211205_IMAP
Record Dates: First submitted 2005-07-11; First posted 2005-07-13 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Cervix Neoplasms
Keywords: Cervix Neoplasms; Vaginal smears; Papillomavirus - Human
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Decision Support Techniques

INTERVENTIONS:
Procedure: HPV DNA testing
Procedure: Conventional management (repeat Pap smear at 6 months)
Procedure: Decision aid with choice of management

SUMMARY:
The study compares the psychosocial outcomes of different management strategies for women with minor atypia (including 'HPV effect') detected on Pap smears: conventional management (a repeat Pap smear at 6 months) versus Human papillomavirus (HPV) DNA testing, a new method proposed for the management of minor atypia and the informed choice of either management supported by a decision aid.

The study examines women's informed preferences for each of these options and compares the psychosocial outcomes in women who are or are not given the choice of management.

HPV DNA testing offers considerable changes to the management of women with minor atypia and there is evidence from the USA which suggests that the use of HPV DNA testing as a triage strategy is effective for women within this group (Solomon et al 2001). The introduction of HPV DNA testing may bring both benefits and harms to women. These harms and benefits are not well understood. Examination of the psychosocial outcomes of HPV DNA testing compared to conventional management and women's preferences for each is needed to guide decisions concerning HPV DNA testing in cervical screening in Australia and also internationally.

DETAILED DESCRIPTION:
Women diagnosed with minor atypia following a routine Pap smear will be randomised into one of the three management arms of the study (a) HPV DNA test, (b) Decision Aid (DA) with choice of management, or (c) a 6 month repeat Pap smear (conventional management). Women who are allocated to the HPV DNA arm and the repeat Pap will receive standard information about their management strategy. Women allocated to the decision aid arm will receive information about HPV DNA testing and 6 month repeat Pap in a decision aid format as an adjunct to usual clinical care and asked to indicate their preference for management. Women in this arm will receive the management strategy of their choice (HPV DNA or repeat Pap). The impact of the Decision Aid will be assessed and psychosocial impact of each management strategy will be followed up over the short, medium and long term.

Management and Clinical outcomes: Data will be collected on the taking and timing of Pap smears, HPV testing and colposcopy as well as findings for each of these tests and any subsequent treatment.

Psychosocial outcomes: Measures will be administered by postal questionnaire at multiple time points across the study. There will be 3 questionnaires: (1) Baseline questionnaire - for all participants recruited into the study; (2) Decision-making evaluation - to assess decision-making in all groups and the impact of the decision aid; (3) Psychosocial impact questionnaire - brief questionnaire (taking approximately 10 minutes to complete) sent at multiple time points to assess the psychosocial impact over time (2 weeks, 3, 6 and 12 months).

Quality of life assessment: Participants will be invited to take part in an interview at 1 month and 12 months post testing (HPV testing or repeat Pap smear) to assess quality of life using standardised validated QOL measures. Interviews will be carried out by an experienced female researcher. Study participants will be given the option to participate in the interview and will be under no obligation to take part if they do not wish to.

ELIGIBILITY:
Inclusion Criteria:

* Women with ONLY the following results on a routine Pap smear:

  * Low grade epithelial abnormality;
  * Minor changes in squamous cell;
  * Minor changes in squamous cells with appearances consistent with Papillomavirus
* Women aged between 18-70 years

Exclusion Criteria:

* Women who are pregnant or planning to become pregnant in the next 12 months
* Women with previous Pap smear abnormality for 2 years.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-01; Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
Psychosocial wellbeing assessed using psychometric scales including (a) global measures of psychological health (STAI, SF36)and (b) measures specific to cervical screening.
Quality of Life (Utility) Assessment two stage standard gamble (SG) technique produces a utility score between 0 and 1.

SECONDARY OUTCOMES:
Clinical outcomes: results of follow-up Pap smear and Colposcopy and HPV testing
Management preference: women's preference for HPV or repeat Pap testing measured by a Decision Aid.
Decision Aid evaluation: Measure the impact of the DA of knowledge, decisional conflict, and satisfaction with decision making

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten McCaffery, PhD, Study Chair — University of Sydney; Les Irwig, PhD, Study Director — University of Sydney; Glenn Salkeld, PhD, Principal Investigator — University of Sydney; Alexandra Barratt, PhD, Principal Investigator — University of Sydney; Kirsten Howard, Masters, Principal Investigator — University of Sydney; Edith Weisberg, Medicine, Principal Investigator — Family Planning Association
Locations (7):
- Australia (7):
  - North Coast Community Health Centre, Port Macquarie, New South Wales
  - Family Planning Association, Sydney, New South Wales
  - Taree Community Health Centre, Taree, New South Wales
  - Illawarra Women's Health Centre, Warilla, New South Wales
  - Family Planning Queensland, Brisbane, Queensland
  - Shine SA, Adelaide, South Australia
  - Family Planning Western Australia, Perth, Western Australia